CLINICAL TRIAL: NCT04497922
Title: Improving Patient Satisfaction Through Information Display Using Virtual White Boards
Brief Title: Virtual White Boards for Patient Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: E-ink corporation (Unknown)
Responsible Party: Principal Investigator, Peter R Chai, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020P002382
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Satisfaction, Patient; Covid19; Emergencies; Satisfaction; Information Disclosure
MeSH Terms: conditions — Patient Satisfaction; COVID-19; Emergencies; Personal Satisfaction | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual in emergency department (Active Comparator): Individuals triaged to a pod in the emergency department without rooms that are fitted with a virtual display screen
  Interventions: Behavioral: Treatment as usual
- Virtual white board (Experimental): Individuals triaged to a pod in the emergency department in a room that is fitted with a virtual display screen
  Interventions: Device: e-ink screen

INTERVENTIONS:
Device: e-ink screen — A virtual display screen developed by e-ink that displays patient status, basic demographics, care team information, pending tests and anticipated disposition
  Arms: Virtual white board
Behavioral: Treatment as usual — Treatment as usual in the emergency department with communication of testing results, imaging and disposition by the primary clinical emergency department team.
  Arms: Treatment as usual in emergency department

SUMMARY:
Communication with patients on their clinical status is important in delivering care in the emergency department. During times of high volume or complex patients, there may be lapses in communicating with patients about their hospital course or plans of action. These miscommunications may be enhanced during the current COVID-19 pandemic as there is minimized in-person interaction with patients in order to conserve personal protective equipment and decrease the risk of disease transmission. This study utilizes a virtual white board to deliver updates to patients about the status of their emergency department stay.

DETAILED DESCRIPTION:
The ultimate goal of this study is to understand the effect of delivering timely information about a patient's emergency department course of their satisfaction surrounding the emergency department stay. The experience of patients in the emergency department has been significantly altered by the COVID-19 pandemic due to decreased in-person encounters, and the use of PPE. Delivering information about their clinical course and expected hospital course is more difficult now given the emphasis on less in-person interaction. In response, the investigators have deployed in collaboration with e-ink, a virtual e-paper white board that can be remotely edited to help display pertinent hospital course information to patients in the emergency department. The investigators will conduct a randomized controlled trial to understand the effect of deploying these white boards on patient satisfaction in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patients in emergency department at Brigham and Women's Hospital
* Triaged to designated emergency department pods outfitted with virtual white board
* Expected emergency department stay of at least four hours
* Able to speak and read english
* Not primary psychiatric complaint

Exclusion Criteria:

* Medically ill or otherwise deemed unable to participate by the study PI and/or treating clinical team.
* Patients admitted to an inpatient bed but boarding in the emergency department over 10 hours.
* Previously participated in the study.
* Has COVID-19 risk flag or confirmed COVID-19 in electronic health record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
emergency department satisfaction: likert scale | 30 minutes after disposition decision for patient
  Satisfaction of overall emergency department stay measured by a 1-5 likert scale, hospital developed question on satisfaction (how satisfied were you with your emergency department stay today?)- higher score is better
Quality of emergency department stay: likert scale | 30 minutes after disposition decision for patient
  Quality of information conveyed to participant (rated on 5 point likert scale on questions about quality of waiting time for test results, staff concern, perceived teamwork in the hospital)

SECONDARY OUTCOMES:
Preference for virtual white board | 30 minutes after disposition decision for patient
  Question on preference for virtual white board compared to a standard emergency department room without a white board (1-4 likert scale, with 4 being strongly prefer white board room)

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Chai, MD MMS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marshall ADA, Hasdianda MA, Miyawaki S, Jambaulikar GD, Cao C, Chen P, Baugh CW, Zhang H, McCabe J, Steinbach L, King S, Friedman J, Su J, Landman AB, Chai PR. A Pilot of Digital Whiteboards for Improving Patient Satisfaction in the Emergency Department: Nonrandomized Controlled Trial. JMIR Form Res. 2023 Mar 21;7:e44725. doi: 10.2196/44725. PMID 36943360